CLINICAL TRIAL: NCT04107779
Title: A Randomized, Open Label, Parallel Group Study in Adult Smokers to Evaluate Changes in Biomarkers of Cigarette Smoke Exposure After Switching Either Exclusively or Partly to Using JUUL Electronic Nicotine Delivery Systems With Two Different Nicotine Concentrations
Brief Title: Changes in Biomarkers of Cigarette Smoke Exposure After Switching Either Exclusively or Partly to JUUL ENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juul Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PROT-00030
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Electronic Cigarette Use; Cigarette Use, Electronic; Tobacco Use; Tobacco Smoking
Keywords: Electronic Nicotine Delivery System; Combustible Cigarettes; Nicotine
MeSH Terms: conditions — Vaping; Tobacco Use; Tobacco Smoking | interventions — Tobacco Products

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Parallel-Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- JUUL 5% Virginia Tobacco ENDS (Experimental): JUUL 5% Virginia Tobacco flavored ENDS product [6 days] in confinement.
  Interventions: Other: Switch from UB of Combustible Cigarette to JUUL 5% Virginia Tobacco ENDS
- JUUL 3% Virginia Tobacco ENDS (Experimental): JUUL 3% Virginia Tobacco flavored ENDS product [6 days] in confinement.
  Interventions: Other: Switch from UB of Combustible Cigarette to JUUL 3% Virginia Tobacco ENDS
- JUUL 5% Mint ENDS (Experimental): JUUL 5% Mint flavored ENDS product [6 days] in confinement.
  Interventions: Other: Switch from UB of Combustible Cigarette to JUUL 5% Mint ENDS
- JUUL 3% Mint ENDS (Experimental): JUUL 3% Mint flavored ENDS product [6 days] in confinement.
  Interventions: Other: Switch from UB of Combustible Cigarette to JUUL 3% Mint ENDS
- JUUL 5% Menthol ENDS (Experimental): JUUL 5% Menthol flavored ENDS product [6 days] in confinement.
  Interventions: Other: Switch from UB of Combustible Cigarette to JUUL 5% Menthol ENDS
- JUUL 3% Menthol ENDS (Experimental): JUUL 3% Menthol flavored ENDS product [6 days] in confinement.
  Interventions: Other: Switch from UB of Combustible Cigarette to JUUL 3% Menthol ENDS
- JUUL 5% Mango ENDS (Experimental): JUUL 5% Mango flavored ENDS product [6 days] in confinement.
  Interventions: Other: Switch from UB of Combustible Cigarette to JUUL 5% Mango ENDS
- JUUL 3% Mango ENDS (Experimental): JUUL 3% Mango flavored ENDS product [6 days] in confinement.
  Interventions: Other: Switch from UB of Combustible Cigarette to JUUL 3% Mango ENDS
- Dual-use of JUUL 5% and UB of Combustible Cigarette (Experimental): JUUL 5% Virginia Tobacco, Mint, Menthol, or Mango flavored ENDS product and usual brand of combustible cigarette [6 days] in confinement.
  Interventions: Other: Switch to Dual-use of JUUL 5% and UB of Combustible Cigarette
- UB of Combustible Cigarette (Active Comparator): Usual brand combustible cigarette [6 days] in confinement.
  Interventions: Other: Usual Brand of cigarettes
- Tobacco/Nicotine Abstention (Other): Smoking abstention (no smoking) [6 days] in confinement.
  Interventions: Other: Tobacco/Nicotine Abstention

INTERVENTIONS:
Other: Switch from UB of Combustible Cigarette to JUUL 5% Virginia Tobacco ENDS — JUUL 5%, ENDS for 6-days in confinement
  Other Names: JUUL
  Arms: JUUL 5% Virginia Tobacco ENDS
Other: Switch from UB of Combustible Cigarette to JUUL 3% Virginia Tobacco ENDS — JUUL 3%, ENDS for 6-days in confinement
  Arms: JUUL 3% Virginia Tobacco ENDS
Other: Switch from UB of Combustible Cigarette to JUUL 5% Mint ENDS — JUUL 5%, ENDS for 6-days in confinement
  Arms: JUUL 5% Mint ENDS
Other: Switch from UB of Combustible Cigarette to JUUL 3% Mint ENDS — JUUL 3%, ENDS for 6-days in confinement
  Arms: JUUL 3% Mint ENDS
Other: Switch from UB of Combustible Cigarette to JUUL 5% Menthol ENDS — JUUL 5%, ENDS for 6-days in confinement
  Arms: JUUL 5% Menthol ENDS
Other: Switch from UB of Combustible Cigarette to JUUL 3% Menthol ENDS — JUUL 3%, ENDS for 6-days in confinement
  Arms: JUUL 3% Menthol ENDS
Other: Switch from UB of Combustible Cigarette to JUUL 5% Mango ENDS — JUUL 5%, ENDS for 6-days in confinement
  Arms: JUUL 5% Mango ENDS
Other: Switch from UB of Combustible Cigarette to JUUL 3% Mango ENDS — JUUL 3%, ENDS for 6-days in confinement
  Arms: JUUL 3% Mango ENDS
Other: Switch to Dual-use of JUUL 5% and UB of Combustible Cigarette — Combination use of JUUL 5% (Virginia Tobacco, Mint, Menthol or Mango flavored) and usual brand combustible cigarettes for 6-days in confinement
  Arms: Dual-use of JUUL 5% and UB of Combustible Cigarette
Other: Tobacco/Nicotine Abstention — No smoking for 6-days in confinement.
  Arms: Tobacco/Nicotine Abstention
Other: Usual Brand of cigarettes — Continue smoking UB for 6-days in confinement.
  Arms: UB of Combustible Cigarette

SUMMARY:
A Randomized, Open Label, Parallel Group Study in Adult Smokers to Evaluate Changes in Biomarkers of Cigarette Smoke Exposure After Switching Either Exclusively or Partly to using JUUL Electronic Nicotine Delivery Systems With Two Different Nicotine Concentrations

DETAILED DESCRIPTION:
Previous studies and data reported in the literature support that Electronic Nicotine Delivery Systems (ENDS) have less toxicant exposure. This study will serve as a clinical evaluation of exclusive-use of selected JUUL ENDS in 2 different nicotine concentrations (5%, 3%), with the purpose of gaining data to support the hypothesis that exclusive-use of JUUL ENDS over the course of 6 days will result in a significant reduction in toxicant exposure compared to combustible cigarettes.

This will be a randomized, open label, parallel group study in adult smokers to be conducted at up to 5 sites in the United States. Changes in Biomarkers of Exposure (BoEs) from baseline when using four JUUL ENDS with 2 different nicotine concentrations (5%, 3%) relative to Usual Brand (UB) of combustible cigarettes and a study group abstaining from any tobacco/nicotine product use will be assessed in this study. JUUL ENDS will be used either exclusively or partially (dual-use), with subjects in the dual-use group using both JUUL 5% ENDS (choice of Virginia Tobacco (VT), Mint, Menthol or Mango flavors) and UB of combustible cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Adult, male or female smoker, 21 to 65 years of age, inclusive, at Screening.
* Has been a smoker for at least 12 months prior to Screening. Brief periods of non-smoking (e.g., up to ~7 consecutive days due to illness, trying to quit, participation in a study where smoking was prohibited) during the 12 months prior to Screening will be permitted at the discretion of the Investigator.
* Currently smokes an average of 10 or more king size or 100s manufactured combustible cigarettes per day, as reported at Screening.
* Cigarettes are the only tobacco product used within (≤) 30 days prior to Screening.
* Has a positive urine cotinine (≥ 200 ng/mL) at Screening.
* Has an exhaled CO > 10 ppm at Screening.
* A female subject of childbearing potential must have been using 1 of the following forms of contraception and agree to continue using it through completion of the study:

  * hormonal (e.g., oral, vaginal ring, transdermal patch, implant, or injection) consistently for at least 3 months prior to Day -2 (Check-in);
  * double barrier method (e.g., condom with spermicide, diaphragm with spermicide) consistently for at least 14 days prior to Day -2 (Check-in);
  * intrauterine device for at least 3 months prior to Day -2 (Check-in);
  * a partner who has been vasectomized for at least 6 months prior to Day -2 (Check-in);
  * abstinence beginning at least 14 days prior to Day -2 (Check-in).
* A female subject of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to Day -2 (Check-in):

  * hysteroscopic sterilization;
  * bilateral tubal ligation or bilateral salpingectomy;
  * hysterectomy;
  * bilateral oophorectomy;
  * Or be postmenopausal with amenorrhea for at least 1 year prior to Day -2 (Check-in) and follicle-stimulating hormone (FSH) levels consistent with postmenopausal status.
* Is willing to comply with the requirements of the study, including a willingness to exclusively use the JUUL products or stop smoking for the duration of the study.
* Provides voluntary consent to participate in this study documented on the signed informed consent form (ICF).

Exclusion Criteria:

* Has a history or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Has a clinically significant abnormal finding on the physical examination, medical history, vital signs, ECG, or clinical laboratory results, in the opinion of the Investigator.
* Has a positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV).
* Has had an acute illness (e.g., upper respiratory infection, viral infection) requiring treatment (including over-the-counter (OTC) remedies) within 14 days prior to Day -2 (Check-in).
* Has a fever (> 100.5°F) at Screening or Day -2 (Check-in).
* Has used prescription or OTC bronchodilator medication (e.g. inhaled or oral βadrenergic agonists) to treat a chronic condition within the 12 months prior to admission;
* Currently has or recently had a bladder or urinary tract infection within 30 days prior to Check-In (Day -2).
* Has a body mass index (BMI) > 40 kg/m2 or < 18 kg/m2 at Screening.
* Has a history of drug or alcohol abuse within 24 months prior to Day -2 (Check-in), as determined by the Investigator
* Has diabetes mellitus, asthma, or chronic obstructive pulmonary disease (COPD).
* Has a systolic blood pressure < 90 mmHg or > 150 mmHg, diastolic blood pressure < 40 mmHg or > 95 mmHg, or heart rate < 40 bpm or > 99 bpm at Screening.
* Has a post-bronchodilator forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC) ratio < 0.7 and FEV1 < 80% of predicted at Screening.
* Has a post-bronchodilator FEV1 increase > 12% and > 200 mL from pre- to post-bronchodilator at Screening.
* Has experienced an allergic reaction following previous e-cigarette use or with exposure to any primary components of the JUUL liquids (benzoic acid, propylene glycol and glycerol).
* Has an estimated creatinine clearance < 70 mL/minute (using the Cockcroft-Gault equation) at Screening.
* Has a positive urine screen for drugs of abuse or positive urine/breath screen for alcohol at Screening or Day -2 (Check-in).
* If female, the subject is pregnant, lactating, or intends to become pregnant during the time period from Screening through the end of study.
* Has used medications known to interact with cytochrome P450 (CYP) 2A6 (including, but not limited to, amiodarone, amlodipine, amobarbital, buprenorphine, clofibrate, clotrimazole, desipramine, disulfiram, entacapone, fenofibrate, isoniazid, ketoconazole, letrozole, methimazole, methoxsalen, metyrapone, miconazole, modafinil, orphenadrine, pentobarbital, phenobarbital, pilocarpine, primidone, propoxyphene, quinidine, rifampicin, rifampin, secobarbital, selegiline, sulconazole, tioconazole, tranylcypromine) within 14 days or 5 half-lives of the drug, whichever is longer, prior to Day -2 (Check-in).
* Has used nicotine-containing products other than manufactured cigarettes (e.g., ENDS, roll-your-own cigarettes, bidis, snuff, nicotine inhaler, pipe, cigar, chewing tobacco, hookah/shisha, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) within 30 days prior to Day -2 (Check-in), except as required per protocol (e.g., the brief product trial at Screening).
* Has a prior history of JUUL product use within (≤) 30 days prior to Screening.
* Has used any prescription smoking cessation treatments, including, but not limited to, varenicline (Chantix®) or buproprion (Zyban®) within 3 months prior to Day -2 (Check-in).
* Is a self-reported puffer (i.e., adult smokers who draw smoke from the cigarette into the mouth and throat but do not inhale).
* Is planning to quit smoking during the study or within 3 months following Day 1, or is postponing a quit attempt in order to participate in the study.
* Negative response (i.e., unwilling to use or unable to tolerate [e.g., experiences Adverse Events during the product trial that will prevent the subjects from continuing to use the JUUL product as judged by the Investigator]) to any of the JUUL products at Screening.
* Has donated plasma within 7 days prior to Day -2 (Check-in).
* Has donated blood or blood products (with the exception of plasma as noted above), has had significant blood loss, or received whole blood or a blood product transfusion within 3 months prior to Day -2 (Check-in).
* Has taken any multivitamin, fish oil or biotin supplements within 48 hours prior to Check-in (Day -2).
* Has consumed any cured meats (e.g., bacon, ham, sausage, corned beef, jerky) or meats cooked at high temperatures (e.g., grilled, fried, smoked or barbecued) within 2 days prior to Check-in (Day -2).
* Has consumed any grapefruit (including grapefruit juice) eggplant or cruciferous vegetables (e.g., cauliflower, cabbage, kale, garden cress, bok choy, broccoli, brussels sprouts and similar green leaf vegetables) within 48 hours prior to Check-in (Day -2).
* Has participated in a previous clinical study for an investigational drug, device, biologic, or tobacco product within 30 days prior to Day -2 (Check-in).
* Is or has a first-degree relative (i.e., parent, sibling, child) who is a current employee of any of the study sites.
* Is or has a first-degree relative (i.e., parent, sibling, child) who is a current employee, shareholder, or is member of the board of directors of JUUL Labs Inc.
* Has previously taken part in, been withdrawn from, or has completed this study.
* Has previously been diagnosed with any form of cancer, except for basal cell or squamous epithelial carcinomas of the skin that have been resected at least 1 year prior to Screening.
* In the opinion of the Investigator, the subject should not participate in this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Primary biomarkers of tobacco exposure measured in urine | 6 days
  Excretion of urine total NNAL, 3-HPMA, MHBMA, and S-PMA will be assessed at baseline and following a 6-day interventional period.
Primary biomarker of tobacco exposure measured in blood | 6 days
  Exposure to carbon monoxide will be assessed through measurement of blood COHb at baseline and following a 6-day interventional period.

SECONDARY OUTCOMES:
Secondary biomarkers of tobacco exposure measured in urine | 6 days
  Excretion of total NNN, total 1-OHP, O-toluidine, 2-NA, 4-ABP, and urine mutagenic activity will be assessed at baseline and following a 6-day interventional period.
Subjective product assessments as measured by the Modified Product Evaluation Scale | 6 days
  Subjective product assessments as measured by responses to the Modified Product Evaluation Scale will be made at baseline and during the interventional period.
Product liking as measured by the Product-Liking Questionnaire visual analog scale | 6 days
  The degree to which subjects like the product will be assessed using the Product-Liking Questionnaire at baseline and during the interventional period.
Urge to smoke as measured by the Urge to Smoke a Cigarette Questionnaire visual analog scale | 6 days
  Urge to smoke as measured by responses to the Urge to Smoke a Cigarette Questionnaire will be assessed at baseline and during the interventional period.
Likelihood of future product use as measured by the Future Intent to Use the Product Questionnaire visual analog scale | 6 days
  Likelihood of future product use as measured by responses to the Future Intent to Use the Product Questionnaire will be made at baseline and during the interventional period.
Daily JUUL product consumption | 6 days
  Daily consumption of the JUUL products as measured by the change in pod weight after use during the interventional period will be reported.
Daily combustible cigarette consumption | 6 days
  Daily consumption of combustible cigarettes as measured by the number of cigarettes smoked per day at baseline and during the interventional period will be reported.
Incidence of adverse events | 6 days
  Safety and tolerability will be assessed by monitoring the incidence of product-use emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rubinstein, MD, Study Director — Juul Labs, Inc.
Locations (5):
- United States (5):
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - St. Louis Clinical Trials, St Louis, Missouri
  - Midwest Clinical Research Center, Dayton, Ohio
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang TW, Asman K, Gentzke AS, Cullen KA, Holder-Hayes E, Reyes-Guzman C, Jamal A, Neff L, King BA. Tobacco Product Use Among Adults - United States, 2017. MMWR Morb Mortal Wkly Rep. 2018 Nov 9;67(44):1225-1232. doi: 10.15585/mmwr.mm6744a2. PMID 30408019
- [Background] U. S. Department of Health and Human Services. The health consequences of smoking - 50 years of progress: A report of the Surgeon General. Department of Health and Human Services, Public Health Service, Office of the Surgeon General. U. S. Government Printing Office, Washington, D. C. (2014)
- [Background] Babb S, Malarcher A, Schauer G, Asman K, Jamal A. Quitting Smoking Among Adults - United States, 2000-2015. MMWR Morb Mortal Wkly Rep. 2017 Jan 6;65(52):1457-1464. doi: 10.15585/mmwr.mm6552a1. PMID 28056007
- [Background] Gottlieb S, Zeller M. A Nicotine-Focused Framework for Public Health. N Engl J Med. 2017 Sep 21;377(12):1111-1114. doi: 10.1056/NEJMp1707409. Epub 2017 Aug 16. No abstract available. PMID 28813211
- [Background] Jensen RP, Luo W, Pankow JF, Strongin RM, Peyton DH. Hidden formaldehyde in e-cigarette aerosols. N Engl J Med. 2015 Jan 22;372(4):392-4. doi: 10.1056/NEJMc1413069. No abstract available. PMID 25607446
- [Background] D'Ruiz CD, Graff DW, Robinson E. Reductions in biomarkers of exposure, impacts on smoking urge and assessment of product use and tolerability in adult smokers following partial or complete substitution of cigarettes with electronic cigarettes. BMC Public Health. 2016 Jul 11;16:543. doi: 10.1186/s12889-016-3236-1. PMID 27401980
- [Background] McNeill A et al. E-cigarettes: An Evidence Update. A report commissioned by Public Health England. Available at: https://www.gov.uk/government/uploads/system/uploads/ attachment_data/file/457102/Ecigarettes_an_evidence_update_A_report_commissioned_by_Public_Health_England_FINAL.pdf (Aug 2015).
- [Background] Polosa R, Morjaria J, Caponnetto P, Caruso M, Strano S, Battaglia E, Russo C. Effect of smoking abstinence and reduction in asthmatic smokers switching to electronic cigarettes: evidence for harm reversal. Int J Environ Res Public Health. 2014 May 8;11(5):4965-77. doi: 10.3390/ijerph110504965. PMID 24814944
- [Background] Tanner JA, Tyndale RF. Variation in CYP2A6 Activity and Personalized Medicine. J Pers Med. 2017 Dec 1;7(4):18. doi: 10.3390/jpm7040018. PMID 29194389
- [Background] HIPAA Privacy Rule. Information for Researchers. De-identifying Protected Health Information Under the Privacy Rule. U.S. Department of Health and Human Services. NIH (Feb 2007). Available at: http://privacyruleandresearch.nih.gov/pr_08.asp#8a.
- [Background] Fagerstrom K. Determinants of tobacco use and renaming the FTND to the Fagerstrom Test for Cigarette Dependence. Nicotine Tob Res. 2012 Jan;14(1):75-8. doi: 10.1093/ntr/ntr137. Epub 2011 Oct 24. No abstract available. PMID 22025545